CLINICAL TRIAL: NCT04998656
Title: Werewolf Flow 50 During ACL Reconstruction: A Randomized Control Trial
Brief Title: Werewolf Flow 50 During ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-2720
Record Dates: First submitted 2021-06-01; First posted 2021-08-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear; Arthrofibrosis of Knee
Keywords: ACL; Anterior Cruciate Ligament; Arthrofibrosis; Knee
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be told whether the Werewolf Flow 50 device was used during their surgery or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Werewolf FLOW 50 Group (Active Comparator): The Werewolf FLOW 50 electrocautery device will be used during surgical treatment for patients assigned to this group.
  Interventions: Device: Werewolf FLOW 50
- Control Group (Placebo Comparator): No electrocautery device will be used during surgical treatment for patients assigned to this group.
  Interventions: Other: Control

INTERVENTIONS:
Device: Werewolf FLOW 50 — Use of Werewolf FLOW 50 electrocautery device during surgical treatment for ACL injury. This device is often used as standard of care when our other standard of care approach (use of no electrocautery device) is not used.
  Arms: Werewolf FLOW 50 Group
Other: Control — Use of no electrocautery device during surgical treatment for ACL injury. This approach is often used as standard of care when our other standard of care approach (use of Werewolf FLOW 50 electrocautery device) is not used.
  Other Names: No Electrocautery Device
  Arms: Control Group

SUMMARY:
The aim of this study is to compare the outcomes, ease of use, and cost of the Werewolf FLOW50 device to the institutional standard of care which is does not include the use of electrocautery devices during anterior cruciate ligament reconstruction (ACLR) surgery in patients 12-18 years of age using a randomized control trial design.

The investigators hypothesize that a lower proportion of participants who undergo ACLR and are randomized to the Werewolf FLOW50 procedure will experience post-operative arthrofibrosis compared to those randomized to standard of care (control group).

DETAILED DESCRIPTION:
The investigators foresee minimal risks to participants. The Werewolf FLOW50 is an FDA approved medical device to be used in the knee joint. he surgeon performing each surgery has used both the Werewolf FLOW50 device (according to FDA-approved indications for use) and no electrocautery device as standard of care during ACL reconstruction surgery.

There is minimal risk associated with the subsequent MRI. Participants may experience slight discomfort from the confined space, flashing lights in their eyes, or temporary warmth/reddening of the skin following MRI. Participants will be informed of these risks and discomforts and pregnant participants or those with any metal and/or electronic devices inside their bodies will not receive the MRI.

There is the risk of unintended disclosure of protected health information (PHI) to individuals outside the research team. To mitigate this risk, data points are entered into a password-protected, HIPAA compliant REDCap database accessible to only the PIs and study personnel. Children's Colorado affiliated and approved study personal will have access to all study information collected at all involved study sites. However, other study sites will only have access to the information collected on patients enrolled at their site. We believe this system will contribute to the protection of PHI. The only PHI collected will be visit dates; all participants will be linked to their information via a unique study identifier.

The PI will periodically review the status of this protocol. Any unanticipated problems will be disclosed to COMIRB [Colorado Multiple Institutional Review Board] within five days with a cover letter detailing the assessment and actions to be taken.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-18 (inclusive) at time of surgery
* Scheduled to undergo ACL reconstruction performed at Children's Hospital Colorado or associated network of care site.

Exclusion Criteria:

* Underlying congenital or musculoskeletal disorders
* Pregnant females, prisoners, and wards of the state
* Persons deemed incompetent and those who have limited decision-making capacity

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Rates of Post-Operative Arthrofibrosis | 1 year post-operative
  Based on post-operative MRIs of the knee, we will compare the rates of post-operative arthrofibrosis between the Werewolf FLOW 50 Group and the Control Group.

SECONDARY OUTCOMES:
Range of Motion | 1 year post-operative
  Based on post-operative clinical examinations, we will compare the knee range of motion between the Werewolf FLOW 50 Group and the Control Group.
Patient Reported Outcomes | 1 year post-operative
  Based on patient reported outcomes (patient surveys) completed pre-operatively and post-operatively, we will compare levels of pain, functionality, overall healing, and quality of life between the Werewolf FLOW 50 Group and the Control Group.
Complications | 1 year post-operative
  We will compare rates of post-operative complications between the Werewolf FLOW 50 Group and the Control Group.

OTHER OUTCOMES:
Procedure Time | Through study completion, an average of 1 year
  After reviewing the operative note in each participant's medical record, we will compare the length of ACL reconstruction procedures between the Werewolf FLOW 50 Group and the Control Group.

CONTACTS AND LOCATIONS:
Overall Officials: Jay C Albright, MD, Principal Investigator — Children's Hospital Colorado
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Main Campus, Aurora, Colorado
  - Children's Hospital Colorado, North Campus, Broomfield, Colorado
  - Children's Hospital Colorado, South Campus, Highlands Ranch, Colorado

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with individuals outside of the authorized study team.

REFERENCES:
- See also: 510(k) Premarket Notification for Werewolf FLOW 50 Device — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K162074